CLINICAL TRIAL: NCT00689364
Title: Retrospective-Prospective Cohort Study Effectiveness of Comprehensive Therapy of TCM to Relieving the Risk of Recurrence and Metastasis for Stage II & III Colorectal Cancer Based on Conventional Western Medicine Therapy
Brief Title: Comprehensive Therapy to Relieving the Risk of Recurrence and Metastasis for Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Collaborators: National Research Centre of Complementary and Alternative Medicine, Norway (Other)
Responsible Party: Xi-Yuan Hospital, China Academy of Chinese Medical Sciences, Department of Oncology, Xi-Yuan Hospital
Other Study IDs: WJB730603
Record Dates: First submitted 2008-05-27; First posted 2008-06-03 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2011-06

CONDITIONS: Colorectal Cancer
Keywords: Cohort Study; Colorectal Cancer; Traditional Chinese Medicine; Risk of recurrence and metastasis
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- CTTCT+CWMT: CTTCM:taking TCM decoction based on syndrome differentiation daily and each dosage is decocted two times for intervention one year with a Chinese patent medicine at least.
  CWMT :with or without chemotherapy/or radiotherapy after the radical operation (R0) (according to the latest NCCN clinical guideline).
- CWMT cohort: CWMT :with or without chemotherapy/or radiotherapy after the radical operation (R0) (according to the latest NCCN clinical guideline).

SUMMARY:
Comprehensive therapy of traditional Chinese medicine (CTTCM) could relieve risk of recurrence and metastasis for stage II & III colorectal cancer, the investigators take this clinical trial with retrospective-prospective cohort study based on previous studies by international multi-center way.

If the study shows a positive result, a pragmatic randomized controlled study with prospective, multi-centre and large-sample design will be given continuously. The aim is to establish recommended programs suggested by CTTCM strategies under conventional Western medicine therapy (CWMT) for stage II & III colorectal cancer.

DETAILED DESCRIPTION:
CTTCM: taking TCM decoction based on syndrome differentiation daily and each dosage is decocted two times for intervention one year with a Chinese patent medicine at least.

CWMT: with or without chemotherapy/or radiotherapy after the radical operation (R0) (according to the latest NCCN clinical guideline).

ELIGIBILITY:
Inclusion Criteria:

* Patient who is diagnosed colorectal cancer by patho& cytologic diagnosis since accepting radical operation within half a year.
* Stage II or III colorectal cancer.
* 18-75 yr.
* Being able to participate and sign the informed consent.

Exclusion Criteria:

* Pregnant woman, Psychotic.
* Patient who put together with other cancer.
* Existed serious complaint and functional disturbance (impairment) with non-tumorous in arch-organ.
* Reactiveness cerebrovascular disease (CVD) .
* Uncontrolled infection and metabolic disease.
* One item of tumor marks is progressed, and it still is progressed when patient recheck.
* Tumor that it is neo-occurred in each organ or pelvic cavity or abdominal cavity without definite patho-quality.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CTTCT plus CWMT cohort in China:160 CWMT cohort in China:160 CWMT cohort in Norway:300
Sampling Method: Non-Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2007-04; Primary Completion 2012-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
The recurrence and metastasis rates for 1、2、3、4 and 5-year. | one year

SECONDARY OUTCOMES:
Survival index: the survival rate for1、2、3、4 and 5-year. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Yang Yufei, doctor, Study Director — Xi-Yuan Hospital, China Academy of Chinese Medical Sciences, China
Locations (1):
- Xi-Yuan Hospital, China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality, China

REFERENCES:
- See also: Related Info — http://www.cctcm.com/